CLINICAL TRIAL: NCT06155071
Title: Effects of 8 Week Plyometric Training on Physical Fitness and Technical Skills of Domestic Cricket Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 014242 Abdul Rehman
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Physical Fitness; Technical Skills
Keywords: Plyometric training; Physical fitness and technical skills; Domestic Cricket players
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Plyometric training) (Experimental)
  Interventions: Other: Plyometric Training
- Group B (Conventional) (Other)
  Interventions: Other: Conventional Exercises

INTERVENTIONS:
Other: Plyometric Training — The group will receive plyometric exercises in a controlled environment. Following Plyometrics would be performed.
  1. Plyo Pushup.
  2. Chest Pass.
  3. Overhead Throw.
  4. Squat jump.
  5. Plyo Step-up.
  6. Cone jumps.
  7. Med Ball drop.
  8. Kneeling Squat jump.
  9. Lateral jump over hurdle.
  10. Overhead throw.
  11. Under hand throws.
  12. Dynamic Rotational Chest pass.
  13. Overhead throw with step.
  Arms: Group A (Plyometric training)
Other: Conventional Exercises — The group will receive conventional exercises in a controlled environment. Following conventional exercises would be performed.
  1. Pushups.
  2. Situps.
  3. Lunges 4.500m running.
  5.Squats
  Arms: Group B (Conventional)

SUMMARY:
This study aims to find the effectiveness of Plyometric training on Physical fitness and Technical skills of Domestic Cricket players. Players would be taken from District Gujrat and a well designed Plyometric training plan will be implied on them for 8 weeks. After the time span the results would be compared to check the effectiveness of the training plan.

DETAILED DESCRIPTION:
Physical improvements have important implications on team sports, as players perform numerous explosive movements like hitting, jumping, turning, sprinting, and changing pace and directions during the match. Cricket requires different roles from each player, and the physical demands vary depending on the format and role.(2) Physiological demands include strength, endurance, speed, agility, power, and flexibility. These physical attributes are essential for effective performance, as they enhance a player's ability to bat, bowl, and field. Good physical fitness enables a player to play at a high level for extended periods of time.

Over the period various training strategies have been used to improve the physical fitness of cricket players. Aerobic training enhances cardiovascular fitness, while resistance training improves maximal strength, vertical jump height, and speed. A combination of weight training and cricket-specific drills are also used to improve both fitness and skills.Physical fitness training can enhance technical skills in cricket players by improving their physical fitness, players is able to execute their technical skills more effectively and with greater precision.

Plyometric training is a type of exercise that involves explosive movements to develop muscular power and enhance physical fitness components.This training is commonly used in many sports activities, including cricket, to improve agility, sprinting, and jumping ability.Research suggests that Ballistic Six plyometric training can increase bowling velocity in medium pace cricket bowlers, leading to improved performance. However, many young cricketers at the domestic level focus only on skill-related fitness, which may not be enough to perform at a high level.While good aerobic capacity is essential for recovery after high-intensity activity, it is anaerobic capacity that ultimately determines success in sports performance.

Components of physical fitness such as Muscular Strength and Power is related to technical skills of cricket as players who have good overall muscular strength and power is able to generate more explosive power in their Bowling and Batting.Agility and speed is enhanced from plyometric training which make the player able to do running effectively during batting and fielding and to change direction instantly as a wicket keeper.Reaction time is also enhanced by plyometric training which have important role in batting and fielding in a cricket game.

However there is no proper or a standard plyometric training program which our domestic cricket players can use as a part of their training plan to enhance their physical fitness and technical skills.Although these plan also affect the technical skill but this aspect lack in the literature.It was hypothesize that game specific plyometric training program may have significant effect on physical fitness as well as technical skills among cricket players.

This study will provide a program of plyometric training which would be quite easy for the players to continue and add in their daily routine, no special equipment would be needed for this and this training program can be done in ground and even players can perform this at their home as well.Effect of this training plan will be beneficial and will enhance not only the physical fitness but will also have effect on the technical skills of our domestic cricket players.

ELIGIBILITY:
Inclusion Criteria:

* domestic cricket players between 15-25 years.
* actively engaged for 1 year

Exclusion Criteria:

* history of trauma/injury in last month

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Aerobic Fitness | 8 weeks
  Yo-Yo test
Endurance | 8 Weeks
  One mile run test.
Flexibilty | 8 weeks
  Sit and reach test
Speed | 8 weeks
  Run a three test
Strength | 8 weeks
  1 rep Max test
Balance | 8 weeks
  Star Excursion balance test
Reaction time | 8 weeks
  Ruler drop test
Bowler accuracy test | 8 weeks
Bowler Speed test | 8 weeks
Throw length test | 8 weeks
Throw accuracy test | 8 weeks
Catching test | 8 weeks
The drop feed | 8 weeks
The bobble feed | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Rehman, Principal Investigator — Riphah International University Islamabad
Locations (1):
- Bestian Cricket Club, Dhok Gujra, Pakistan

IPD SHARING:
Plan to Share IPD: No